CLINICAL TRIAL: NCT03999879
Title: Neuroenergetic Adaptations in Alzheimer's Disease: Implications on Amyloid Burden and Cognition.
Brief Title: PhosphoRus, Proton Imaging and Amyloid BuRdEn (PREPARE) ON AMYLOID BURDEN AND COGNITION
Acronym: PREPARE
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 18-01919
Record Dates: First submitted 2019-06-25; First posted 2019-06-27 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cognitively Normal: having 30 participants with normal cognition
  Interventions: Diagnostic Test: Measure of OxPhos upregulation; Diagnostic Test: lactate (measured with 1H-MRSI)
- Amnesic MCI: aMCI Group having 15 participants with a CDR of 0.5-1 and a Mini-Mental State Examination (MMSE) of 20-25.
  Interventions: Diagnostic Test: Measure of OxPhos upregulation; Diagnostic Test: lactate (measured with 1H-MRSI)

INTERVENTIONS:
Diagnostic Test: Measure of OxPhos upregulation — OxPhos upregulation [i.e., lower phosphocreatine (PCr)-to-ATP ratio levels] in the PET AG mask. PIB+ NL subjects will show OxPhos downregulation (i.e. increased PCr/ATP ratio that indicate the presence of metabolically inert PCr that cannot be used as ATP) when compared to PIB- NL subjects in the PETAG mask
Diagnostic Test: lactate (measured with 1H-MRSI) — PIB+ NL subjects will show increased levels of lactate (measured with 1H-MRSI) when compared to PIB- NL subjects in the PETAG mask.

SUMMARY:
Normal cells primarily produce energy with the help of the "mitochondria". These "small organs" are also called the "powerhouses of the cell" turn the sugars, fats and proteins that is eaten into forms of chemical energy that the body can use to carry on living. This process is called oxidative phosphorylation. In addition to the help from the mitochondria and oxidative phosphorylation, most cells can produce energy by lactic acid fermentation. This process is less energy efficient but faster and used by the brain, muscle or other organs under specific circumstances and energy demands, even in the presence of abundant oxygen. It is also called aerobic glycolysis. Aerobic glycolysis and oxidative phosphorylation are the two major mechanisms involved in brain energetics.

DETAILED DESCRIPTION:
The consequences of Alzheimer's disease (AD) (deposition of amyloid plaques and neurofibrillary tangles) are known. The cause of these deposition of proteins is not. Some scientist argue that an increase in oxidative phosphorylation activity and a lack of ability to shift to aerobic glycolysis are the underlying source of these changes. The purpose of this study is to test whether there is a correlation between neuroenergetic levels of aerobic glycolysis/oxidative phosphorylation and risk for Alzheimer's disease. The study will examine these neuroenergetic adaptations in a group of 15 elderly participants (age range: 70-85 y/o) with amnestic mild cognitive impairment (aMCI) and 30 cognitively normal controls (NL). Multimodal (MR/PET) and multinuclear (31P/1H) neuroimaging will allow us to gain access to a uniquely comprehensive and highly consistent view of neuroenergetic adaptations in both the clinical and preclinical stages of Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* NL Group: Adults (male and female) aged >70 years in overall excellent health with normal cognition (CDR=0), and at least high school graduate level education.
* aMCI Group: Adults (male and female) aged >70 years, Clinical Dementia Rating (CDR)= 0.5 - 1 and Mini-Mental State Examination (MMSE): 20-25
* English as first language or demonstrated proficiency in English for non-native speakers

Exclusion Criteria:

* Any tumor, stroke, or trauma that would result in abnormal radiological findings History of bipolar disorder, schizophrenia, intellectual disability or substance abuse MRI scanner contraindications

Ages: 70 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Adults (male and female) aged >70 years in overall excellent health with normal cognition (CDR=0), and at least high school graduate level education.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2023-02-24 (Actual); Study Completion 2023-02-24 (Actual)

PRIMARY OUTCOMES:
(PCr)-to-ATP ratio levels | 1 Month
  These 31P-MRSI data will differentiate PiB+ aMCI individuals from PiB+ NL individuals.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Brown, MD, Principal Investigator — New York Langone Medical Center
Locations (1):
- New York University School of Medicine, New York, New York, United States

DOCUMENTS (1):
  • Informed Consent Form (2022-05-09): https://cdn.clinicaltrials.gov/large-docs/79/NCT03999879/ICF_000.pdf